CLINICAL TRIAL: NCT07078929
Title: Safety and Preliminary Efficacy of CD19 With IL-7 Receptor Alpha Signaling Chimeric Antigen Receptor T Cell (CMD63) in Relapse and Refractory Pediatric B-cell Acute Lymphoblastic Leukemia
Brief Title: Phase I Clinical Trial of CMD63 CAR T Cell in Children With Acute Lymphoblastic Leukemia
Acronym: CMD63
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMD63-ALL-2025; Chulalongkorn University (Other: Chulalongkorn University)
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Relapse B Acute Lymphoblastic Leukemia; Refactory Childhood Acute Lymphoblastic Leukemia
Keywords: CAR T cell; CD19; IL-7 receptor alpha; Chimeric antigen receptor T cell; Adoptive cellular therapy; B-cell acute lymphoblastic leukemia
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Intervention Model Description: 3+3 dose escalation study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19 IL-7Ra CAR T cell in B-cell acute lymphoblastic leukemia (Experimental): CD19-specific chimeric antigen receptor (CAR) T cell with IL-7 receptor alpha signaling Dose level: 0.5x10e6 cells/kg, 1x10e6 cells/kg
  Interventions: Biological: CD19-IL7Ra CAR-T cells

INTERVENTIONS:
Biological: CD19-IL7Ra CAR-T cells — Autologous T cells lentiviral transduced to express a CD19-specific chimeric antigen receptor (CAR) with the addition of an IL-7 receptor alpha signaling domain, administered via central venous access catheter after lymphodepletion

SUMMARY:
A Phase 1 clinical trial to evaluate the safety and early efficacy of CAR T-cells with IL-7Rα signaling targeting CD19 in children with relapsed and refractory B-cell acute lymphoblastic leukemia after complete standard treatments.

DETAILED DESCRIPTION:
Hematological cancers are a significant public health problem in Thailand. Currently, treatment outcomes for patients with B-cell leukemia using standard chemotherapy regimens show satisfactory disease control and survival rates. However, patients with relapsed or refractory disease have very limited treatment options, as the chance of achieving remission through chemotherapy or targeted therapies before bone marrow transplantation is less than 20%. Once patients experience relapse or become refractory to treatment, their chance of surviving more than one year is extremely low. Therefore, developing new treatments for relapsed or refractory B-cell leukemia is urgently needed to provide additional treatment options, increase response rates, and improve survival outcomes in these patients.

Phase 1 to Phase 3 clinical research studies worldwide have demonstrated that treating patients with relapsed or refractory B-cell leukemia using the patients' own genetically modified T cells that specifically target B-cell leukemia and lymphoma cells can control the disease in 70-90% of B-cell leukemia patients. Approximately 50-60% of patients survive without disease recurrence for more than one year after treatment, with manageable side effects.

For these reasons, this research project aims to study the safety of treating Thai pediatric patients with relapsed or refractory B-cell leukemia using the patients' own T cells that have been genetically modified to become chimeric antigen receptor T cells specifically targeting proteins on the surface of leukemia cells. This research is being conducted for the first time in Thai pediatric patients. The research team expects this treatment to be highly safe and effective in controlling B-cell leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have relapsed, or refractory ALL treated with at least one lines of therapy. Disease must have either progressed after the last regimen or presented failure to achieve complete remission with the last regimen.

   - Participant with Philadelphia Chromosome positive ALL are eligible if the progressed, had stable disease or relapsed after one line of therapy including tyrosine kinase inhibitors (TKIs)
2. The participant's disease must be CD19 positive either by immunohistochemistry or flow cytometry analysis
3. Age 1 - 18 years
4. Sex: Male or Female
5. Performance status: Lansky or Karnofsky score greater than or equal to 50
6. Normal organ function:

   * AST (SGOT) less 5 times the upper limit of normal (ULN)
   * ALT (SGPT) less 5 times the upper limit of normal (ULN)
   * Total bilirubin less 3 times the upper limit of normal (ULN)
   * Creatinine less 5 times the upper limit of normal (ULN)
   * SpO2 room air greater than or equal to 90%
7. Prior therapy wash-out before planned leukapheresis 7.1 Greater than or equal to 7 days post last chemotherapy/biologic therapy administration 7.2 Three half-lives or 30 days, whichever is shorter after the last dose of antitumor antibody therapy 7.3 At least 30 days from most recent cellular infusion 7.4 All systemically administered corticosteroid treatment therapy must be stable or decreasing within 1 week prior to enrollment with a maximum of 0.5 mg/day dose of methylprednisolone. Corticosteroid physiologic replacement therapy is allowed
8. Participants and/or care givers must have the ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

1. Active GVHD that required systemic immunosuppressant with 4 weeks of enrollment
2. History of active malignancy other than non-melanoma skin cancer and carcinoma in situ (e.g. cervix, bladder, breast).
3. Participants with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, pulmonary abnormalities, Graft Versus Host Disease or psychiatric illness/social situations that would limit compliance with study requirements.
4. Pregnant or breastfeeding women are excluded from this study because CAR-T cell therapy may be associated with potential for teratogenic or abortifacient effect. Women of child bearing potential must have negative serum pregnancy test. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of mother with CAR-T cells, breast feeding should be discontinued. These potential risks may also apply to other agents used in this study. Participants of child-bearing or child-fathering potential must be willing to practice birth control from the time of enrollment on this study and for four months after receiving CAR-T cell infusion.
5. Evidence of myelodysplasia or cytogenetic abnormality indicative of myelodysplasia on any bone marrow biopsy prior to initiation of therapy.
6. Serologic status reflecting active HIV, hepatitis B or C infection. Participants that are positive for hepatitis B core antibody, hepatitis B surface antigen or hepatitis C antibody must have negative PCR prior to enrollment.
7. Participants who have a history of anaphylactic reaction to albumin.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of CD19-IL7Ra CAR T-cells infusion in B-cell acute lymphoblastic leukemia patients. | 7 days, 14 days, 21 days, 30 days, 60 days, 90 days, 6 months and 12 months after CD19-IL7Ra CAR-T cell infusion
  The incidence of adverse events assessed by the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 5.0

SECONDARY OUTCOMES:
The overall response rate of B-cell acute lymphoblastic leukemia | 30 days, 60 days, 90 days, 6 months and 12 months after CD19-IL7Ra CAR-T cell infusion
  The overall response rate will be assessed using standard response criteria for acute lymphoblastic leukemia patients through a combination of clinical, hematologic, and molecular assessments. The response categories are Minimal Residual Disease (MRD), Complete Response (CR), Complete Response with Incomplete Count Recovery (CRi), Stable Disease (SD), and Progressive Disease (PD).

OTHER OUTCOMES:
Persistence of anti-CD19 CAR-T cell in peripheral blood | 7 days, 14 days, 21 days, 30 days, 60 days, 90 days, 6 months and 12 months after CD19-IL7Ra CAR-T cell infusion
  Persistence of anti-CD19 CAR-T cell in peripheral blood of leukemia patients measuring by flow cytometry and qPCR.
Serum cytokine level measurement | 7 days, 14 days, 21 days and 30 days after CD19-IL7Ra CAR-T cell infusion
  Serum cytokine level measurement including IL-2,IL-4, IL-6, IL-10, TNF-alpha and IFN-gamma before and after CD19-IL7Ra CAR T-cell infusion

CONTACTS AND LOCATIONS:
Overall Officials: Kanhatai Chiengthong, MD, Principal Investigator — King Chulalongkorn Memorial Hospital
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Pathumwan, Thailand

IPD SHARING:
Plan to Share IPD: No